CLINICAL TRIAL: NCT06836466
Title: Physicians' Awareness of ECG Abnormalities Linked to Acute Ischemic Chest Pain; A Survey Study
Brief Title: Physicians' Awareness of ECG Abnormalities Linked to Acute Ischemic Chest Pain
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ezzat Nasreddin, Lecturer of Emergency and Traumatology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR955/11/24
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Physicians; Awareness; ECG Abnormalities; Acute Ischemic Chest Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All physicians are subjected to 10 ECGs Surves
  Interventions: Other: Google Form-based questionnaire

INTERVENTIONS:
Other: Google Form-based questionnaire — All participants will consent to submit an anonymous Google Form-based questionnaire. The designed questionnaire includes introductory personal, academic, and work experience data about the physicians as gender, age, current specialty, workplace, highest achieved medical-academic or training degree, and number of years of postgraduate clinical work experience.

SUMMARY:
This study aims to investigate physicians' awareness regarding patients presenting with potential acute ischemic chest pain. It focuses on various electrocardiogram (ECG) patterns requiring prompt catheter lab activation for reperfusion therapy alongside other ECG mimics that may lead to false catheter lab activations.

DETAILED DESCRIPTION:
Chest pain is the second most common complaint in adult emergency department (ED) patients in the United States. Most visits result in a diagnosis of noncardiac chest pain and approximately half in nonspecific chest pain. Roughly 6% are ultimately diagnosed with a life-threatening condition, which is overwhelmingly (>90%) acute coronary syndrome (ACS).

The term acute coronary syndrome (ACS) is applied to patients in whom there is a suspicion or confirmation of acute myocardial ischemia or infarction. ST-elevation myocardial infarction (STEMI), Non-ST-elevation MI (NSTEMI), and unstable angina are the three traditional types of ACS.

ELIGIBILITY:
Inclusion Criteria:

* Age from 25 to 65 years.
* Both sexes.
* Physicians who treat patients with possible acute chest pain.

Exclusion Criteria:

- Participants who failed to complete the survey questions.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive sample of 500 physicians who treat patients with possible acute ischemic chest pain will be the subject of this cross-sectional survey study. These doctors will include emergency physicians, cardiologists, internal medicine/acute medicine specialists, general practice or family physicians, anesthesiologists, and intensive care physicians of both sexes, with varying degrees of experience and post-graduate clinical training, from all over the world.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Physicians' Awareness | At time of online survey (Up to 2 months)
  Physicians' awareness is measured by a numerical score of 0 to 10, depending on the electrocardiogram (ECG) pattern survey. 0 means (least recognition of ECG pattern) and 10 (high recognition of ECG pattern)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.